CLINICAL TRIAL: NCT03405883
Title: Comparative Analysis of the Uterine Microbiome in Women with Repeated Implantation Failure and Normal Fertile Women
Brief Title: Uterine Microbiome in Women with Repeated Implantation Failure and Normal Fertile Women
Status: Completed | Type: Observational
Sponsor: University Hospital, Ghent (Other)
Collaborators: University Ghent (Other)
Responsible Party: Sponsor
Other Study IDs: BE670201733152
Record Dates: First submitted 2018-01-12; First posted 2018-01-23 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Repeated Implantation Failure; Normal Fertile

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Microbiome analysis using 16S ribosomal RNA sequencing
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- RIF (women with repeated implantation failure): Transfer of at least 5 good quality embryos in IVF or ICSI cycles, without achieving pregnancy
  Interventions: Other: Vaginal swab + endometrial biopsy
- NF (normal fertile women): Spontaneous conception or conception after max 9 IUI cycles
  Interventions: Other: Vaginal swab + endometrial biopsy

INTERVENTIONS:
Other: Vaginal swab + endometrial biopsy — In the midluteal phase of the cycle, a vaginal swab (E swab) and endometrial biopsy (TAO brush) will be obtained.

SUMMARY:
Characterization of the uterine microbiome in women with repeated implantation failure as well as in normal fertile women.

DETAILED DESCRIPTION:
In the midluteal phase of the cycle, a vaginal swab and endometrial biopsy will be obtained.

ELIGIBILITY:
Inclusion Criteria:

* Women between their 18th and 40th birthdays (max 39 years and 364 days at the day of signing the informed consent)
* Able to understand, read and speak Dutch and hence to provide written and oral informed consent
* Negative serological tests for human immunodeficiency virus (HIV), hepatitis B virus (HBV), hepatitis C virus (HCV), Rapid plasma reagin (RPR) for syphilis

Exclusion Criteria:

* Hormonal contraception in current cycle
* Presence of intra-uterine device
* Antibiotic treatment in the current cycle

Ages: 18 Years to 39 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: * For RIF women: absence of pregnancy after transfer of in total 5 embryos of high quality embryos
  * For NF women: live birth after spontaneous conception or IUI (max 9x)
Sampling Method: Non-Probability Sample
Enrollment: 13 (Actual)
Dates: Start 2018-01-01 (Actual); Primary Completion 2018-12-31 (Actual); Study Completion 2018-12-31 (Actual)

PRIMARY OUTCOMES:
Midluteal uterine microbiome profile | 1 week
  Descriptive analysis of the uterine microbiome present

SECONDARY OUTCOMES:
Midluteal vaginal microbiome profile | 1 week
  Descriptive analysis of the vaginal microbiome present (quality control of endometrial sampling)

CONTACTS AND LOCATIONS:
Overall Officials: Hans Verstraelen, MD, PhD, Principal Investigator — University Hospital, Ghent
Locations (1):
- Ghent University Hospital, Ghent, Belgium

IPD SHARING:
Plan to Share IPD: Undecided